CLINICAL TRIAL: NCT00478140
Title: A Phase II Study Trastuzumab (NSC 688097) in Her2/Neu Positive Cancer of the Gallbladder or Biliary Tract (NCI 7756)
Brief Title: Trastuzumab in Treating Patients With Locally Advanced or Metastatic Gallbladder Cancer or Bile Duct Cancer That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00217; 2006-0851; N01CM62202 (NIH)
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Adenocarcinoma of the Extrahepatic Bile Duct; Adenocarcinoma of the Gallbladder; Malignant Neoplasm; Recurrent Extrahepatic Bile Duct Cancer; Recurrent Gallbladder Cancer; Unresectable Extrahepatic Bile Duct Cancer; Unresectable Gallbladder Cancer
MeSH Terms: conditions — Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab (Experimental): Participants receive trastuzumab loading dose 8 mg/kg intravenous (IV) over 30-90 minutes on day 1 and subsequent maintenance doses of 6 mg/kg over 90 minutes then every 30 minutes starting at the third dose. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: trastuzumab — For HER-2/neu positive biopsies, trastuzumab was administered intravenously, once every 3 weeks, at a loading first dose at 8 mg/kg over 90 minutes, and subsequent maintenance doses of 6 mg/kg over 90 minutes then every 30 minutes starting at the third dose.
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well trastuzumab works in treating patients with locally advanced or metastatic gallbladder cancer or bile duct cancer that cannot be removed by surgery. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the objective response rate and duration of objective response in patients with HER2/neu-positive advanced gallbladder or biliary tract cancer treated with trastuzumab (Herceptin).

SECONDARY OBJECTIVES:

I. Assess the safety and tolerability of this drug in these patients. II. Assess the progression-free survival and overall survival of patients treated with this drug.

OUTLINE:

Patients receive trastuzumab intravenously over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Criteria:

* Adenocarcinoma of the gallbladder
* Recurrent extrahepatic bile duct cancer
* Recurrent gallbladder cancer
* Unresectable extrahepatic bile duct cancer
* Adenocarcinoma of the extrahepatic bile duct
* Unresectable gallbladder cancer
* Prior surgery and radiotherapy allowed
* At least 28 days since prior chemotherapy (6 weeks for nitrosoureas and mitomycin C) and recovered
* No other concurrent investigational agents, chemotherapy, radiotherapy, or hormonal therapy
* Concurrent hormones administered for nondisease-related conditions (e.g., insulin for diabetes) allowed
* No concurrent corticosteroids or anticonvulsants
* Concurrent steroids administered for antiemesis, adrenal failure, or septic shock allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Histologically or cytologically confirmed adenocarcinoma of the gallbladder or bile duct, meeting all of the following criteria: locally advanced or metastatic disease that is unresectable
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques or >= 10 mm by spiral computed tomography (CT) scan
* Tumor that recurs within a previously irradiated field is considered measurable disease if recurrence is documented and measurable by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Tumor must be Her2/neu positive by Fluorescence in situ hybridization (FISH)testing
* No symptomatic brain metastases
* The Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Fertile patients must use effective contraception prior to, during, and for >= 3 months after completion of study treatment
* Creatinine =< 2 times upper limits of normal (ULN) OR creatinine clearance >= 60 mL/min
* No other active malignancy
* Left Ventricular Ejection Fraction (LVEF) >= 50%
* No concurrent uncontrolled illness
* No ongoing or active infection requiring systemic IV antibiotics on day 1 of treatment
* No symptomatic New York Heart Association class III-IV congestive heart failure
* No unstable angina pectoris
* No unstable cardiac arrhythmia requiring medication
* No more than 1 prior systemic chemotherapy regimen
* White Blood Count (WBC) >= 3,000/mm^3
* Platelet count >= 40,000/mm^3
* Bilirubin =< 4 mg/dL
* Aspartate aminotransferase and alanine aminotransferase (AST and ALT) =< 5 times upper limit of normal (ULN)
* Not pregnant or nursing
* Negative pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kaseb, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - The University of Texas (UT) MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 30, 2007 to June 15, 2009. All recruitment done in medical clinics.
Pre-assignment Details: Of the 53 participants pre-screened only four participants were enrolled in the study.
Groups:
- Trastuzumab: Trastuzumab loading dose 8 mg/kg intravenous (IV) over 30-90 minutes on day 1 and subsequent maintenance doses of 6 mg/kg over 90 minutes then every 30 minutes starting at the third dose. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Trastuzumab
Started | 4
Completed | 3
Not Completed | 1
Not completed — Clinical Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 52 [38 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete and Partial Response)
Description: Response assessed using imaging-based evaluation at baseline then following single agent trastuzumab administered over 21 day cycle, re-staging done following 2 cycles. Response Evaluation Criteria in Solid Tumors defined as Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in sum of longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Baseline to 63 days or until disease progression
Population: Only those participants who had measurable disease present at baseline, received at least one cycle of therapy, and had disease re-evaluated considered evaluable for response; therefore one participant was inevaluable.
Measure: Number; unit: participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 3
participants
  Complete Response | 1
  Partial Response | 0
  Progressive Disease | 1
  Stable Disease | 1

2. Secondary Outcome: Disease Control Rate
Description: Percentage of participants who have achieved complete response, partial response and stable disease
Time Frame: Up to 3.5 years
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 3
percentage of participants | 67

3. Secondary Outcome: Number of Participant With Toxicity Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: Participant toxicity for study as assessed using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 reported in Results Adverse Event Reporting of record.
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 3
participants | 3

4. Secondary Outcome: Overall Survival
Description: Length of time from date of starting treatment that participants are still alive
Time Frame: Up to 3.5 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Trastuzumab
Number analyzed (Participants) | 3
weeks | 65 [9.4 to 127]

ADVERSE EVENTS:
Time Frame: 2 years and 9 months
Arm/Group | Trastuzumab
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=4)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Allergic reaction (Immune system disorders) | 2
Allergic rhinitis (Immune system disorders) | 2
Anorexia (Gastrointestinal disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Ascites (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 4
Gastrointestinal disorders (Gastrointestinal disorders) | 2
Insomnia (General disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Weight loss (Investigations) | 2
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 2
Blood bilirubin increased (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Creatinine increased (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysgeusia (Gastrointestinal disorders) | 1
Fever (Infections and infestations) | 1
Headache (General disorders) | 3
Hyperkalemia (Blood and lymphatic system disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Mucositis oral (Respiratory, thoracic and mediastinal disorders) | 1
Myalgia (Cardiac disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Chills (Investigations) | 2
Cystitis noninfective (Renal and urinary disorders) | 1
Hematuria (Blood and lymphatic system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Hyperhidrosis (Nervous system disorders) | 1
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less